CLINICAL TRIAL: NCT05535179
Title: The Application of Gargle Containing Honeysuckle and Semen Oroxyli to Reduce the Pain and Complications After Uvulopalatopharyngoplasty
Brief Title: Effect of Gargle Containing Honeysuckle and Semen Oroxyli
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hubei Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Zhongyi Miao, Director, Hubei Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HubeiHTCM 001
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Obstructive Sleep Apnea; Complication; Pain
MeSH Terms: conditions — Sleep Apnea, Obstructive; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental)
  Interventions: Drug: honeysuckle and semen oroxyli solution
- control group (No Intervention)

INTERVENTIONS:
Drug: honeysuckle and semen oroxyli solution — The patients in the treatment group were instructed to gargle the solution containing honeysuckle and semen oroxyli (25 mL) four times a day for 2 weeks.
  Arms: treatment group

SUMMARY:
Surgery All patients included in this study underwent UPPP under general anesthesia with a low-temperature plasma ablation apparatus (PLA-600; Zhongyuan Medical Equipment Co., Ltd.; Shandong, China). Briefly, the surgery was carried out under general anesthesia using a nasal cannula. A 70# low-temperature plasma cutter head was used to perform bilateral epicapsular ablation of the tonsils. Inverted "U" incisions were made on the bilateral soft palate respectively, and the 70# cutter head progressively melted the adipose tissue and other soft tissues in the the veli palatine region. Subsequently, a 55# low-temperature plasma cutter head was used to perform perforation and ablation from between the two mucosal layers of the soft palate to the direction of the hard palate, with 2-3 holes on each side, and each ablation time was 8-12 s.

Treatments Patients in both the 2 groups received amoxicillin sodium suspension every 8 hours for 7 days after UPPP. Except for these drugs, patients in the treatment group were instructed to gargle the suspension solution containing honeysuckle and semen oroxyli (25 mL) for 5 minutes. The solution was given 4 times a day for 2 weeks. The patients in the control group were instructed to gargle normal saline (25 mL) at the same schedule. No NSAIDs were administered unless requested by the patient.

Data collection The post-operative resting throat pain and swallowing throat pain were evaluated at 0 week (12 hours after surgery), 1 week and 2 weeks after UPPP by the patients themselves using a visual analog scale (VAS) based on a linear scale from 0 to 10, where 0 represented an absence of pain and 10 represented maximal pain. Then, the changes of scores from week 0 to week 2 between the 2 groups were compared. The VAS scores related to patient comfort level were also evaluated by patients themselves, with 0 representing very much worse and 10 very much comfort. Furthermore, the researchers who were blinded to the therapeutic regimens evaluated the improvement in postoperative pain of patients within the 2-week postoperative period based on the clinical global impression of improvement (CGI-I score) questionnaire. In this questionnaire, the researchers used a seven-point scale from 1 (very much improved) to 7 (very much worse) to rate the improvement of body pain of the patients (10).

The post-operative complications, such as wound infection and wound bleeding, were collected and analyzed. The baseline characteristics of the patients in 2 groups including age, gender, body mass index (BMI), OSA severity, American Society of Anesthesiologist (ASA) classification and pre-operative complications were also collected. The venous blood was collected at 12 h and 1 week after operation to detect the levels of hs-CRP, hemoglobin, neutrophil% and white blood cell count (WBC).

Statistical analysis The data in this study were analyzed by the SPSS software (version 22.0). Normal distribution quantitative data were described as mean ± SD. The difference between groups were compared by the Student's t test. Non-normal distribution quantitative data were described as median with range and compared with Mann-Whitney U test. Categorical data were described as numbers and percentages and compared using the Chi-square test or Fisher's exact test. P < 0.05 was considered as statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had undergone elective UPPP during the period of April 2019 to January 2022

Exclusion Criteria:

* patients with a history of systemic diseases such as severe cardiac and/or pulmonary disorders;
* patients who were unable to cooperate with evaluations;
* patients with severe diabetes;
* patients who had underwent other surgeries in the last 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Comparison of resting throat pain in two groups | 1 week and 2 weeks after UPPP
  For resting throat pain at 1 week and 2 weeks after UPPP, the VAS scores of the treatment group were much lower than those of the control group (P = 0.033 and P = 0.031, respectively, Table 2). However, the VAS scores for resting throat pain measured at 12 h after UPPP were not significantly different between the 2 groups (P = 0.465).
Comparison of swallowing throat pain in two groups | 12 h, 1 week and 2 weeks after surgery
  For swallowing throat pain, treatment group had much lower VAS scores than control group at 2 weeks after surgery (P < 0.001). But the 2 groups had similar VAS scores for swallowing throat pain at 12 h and 1 week after surgery (P = 0.414 and 0.732, respectively)
Comparison of changes in VAS scores between the two groupd for both resting and swallowing throat pain | week 0 to week 2
  The changes of VAS scores for both resting and swallowing throat pain from week 0 to week 2 were significantly higher in treatment group than in control group (P < 0.001 and P = 0.005, respectively).
Comparison of GGI-I score in two groups | week 0 to week 2
  The treatment group performed a lower GGI-I score than control group (P < 0.001)
Comparison of total complication rates in two groups | 2 weeks after surgery
  No deaths occurred within the 2-week postoperative period. The total complication rates between the 2 groups was not significantly different (P = 0.071)
Comparison of post-operative wound infection or wound bleeding between two groups | 2 weeks after surgery
  Although the treatment group had less numbers of patients with post-operative wound infection or wound bleeding, the difference between the 2 groups was not statistically significant.
Comprision of the levels of hs-CRP, hemoglobin, neutrophil% and WBC between the 2 groups | 12 h after surgery and 1 week after sugery
  The levels of hs-CRP, hemoglobin, neutrophil% and WBC between the 2 groups at 12 h after surgery were not significantly different. One week after operation, the levels of hs-CRP, Hemoglobin, and WBC in the treatment group were significantly lower than those in the control group (P<0.05).

CONTACTS AND LOCATIONS:
Locations (1):
- Hebei Hospital of traditional Chinese Medicine, Shijiazhuang, Hebei, China